CLINICAL TRIAL: NCT02602743
Title: Propofol-Ketamine vs Remifentanyl-Ketamine for Sedation in Pediatric Patients Undergoing Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Specialist Doctor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRK01
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Delayed Emergence From Anesthesia
Keywords: sedation; remifentanyl; pediatric patient; colonoscopy
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Remifentanil; Propofol; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanyl, ketamine (Experimental): Experimental:Remifentanyl and ketamine Remifentanyl vial 2 mg, Ketamine vial 500mg/10 mlt by intravenous. 2 mg/kg ketamine and 0,25 µg/kg remifentanyl will be administered for induction in 1 minute. Then 0,1 µg/kg/h remifentanyl infusion will be started.
  Interventions: Drug: Remifentanyl; Drug: Ketamine
- propofol, ketamine (Active Comparator): Active comparator:Propofol and ketamine Propofol injectable emulsion vial 200 mg/20 mlt, Ketamine vial 500mg/10 mlt by intravenous.
  2 mg/kg ketamine and 1 mg/kg propofol will be administered for induction and then 1 mg/kg/h propofol infusion will be started.
  Interventions: Drug: Propofol; Drug: Ketamine

INTERVENTIONS:
Drug: Remifentanyl — 0,25 µg/kg remifentanyl will be administered for induction in 1 minute. Then 0,1 µg/kg/h remifentanyl infusion will be started.
  Other Names: Ultiva
  Arms: remifentanyl, ketamine
Drug: Propofol — 1 mg/kg propofol will be administered for induction and then 1 mg/kg/h propofol infusion will be started.
  Other Names: Pofol
  Arms: propofol, ketamine
Drug: Ketamine — 2 mg/kg ketamine will be administered for induction in 1 minute.
  Other Names: Ketalar

SUMMARY:
Ketamine and propofol have been used most frequently agents and remifentanil is used with increasing frequency in recent years. Investigators will compare ketamine-propofol and ketamine-remifentanyl effects on drug consumption, respiration, hemodynamics and recovery in pediatric colonoscopy patients. Our study is a prospective, randomized comparison of ketamine-propofol and remifentanyl-propofol for sedation in pediatric patients during elective colonoscopy. ASA I-II, 2-16 years old, seventy children will be included in the study after ethics committee approval and written informed consent from the parents. Children with cardiovascular, cerebral, pulmonary, renal and hepatic diseases will be excluded from the study. Group I (RK); 2 mg/kg ketamine and 0,25 µg/kg remifentanyl will be administered for induction in 1 minute.Then 0,1 µg/kg/h remifentanyl infusion will be started.

Group II (PK); 2 mg/kg ketamine and 1 mg/kg propofol will be administered for induction and then 1 mg/kg/h propofol infusion will be started. In case of movement, crying, heart rate and systolic blood pressure more than 20% increase from baseline; 0.05 to 0.1 mg / kg of remifentanil will be administered in group I, 0.5-1 mg / kg will be administered propofol in group II. Not enough that case 0.5-1 mg / kg of ketamine will be applied.

The anesthesiologist will continue monitoring after completion of colonoscopy until recovery of full consciousness. A Steward recovery score of 7 will be defined as the end of the recovery time.

DETAILED DESCRIPTION:
Optimal drug combinations for sedation and analgesia for the diagnosis and treatment of interventional procedures performed in pediatric patients still continue to be the main subject of many scientific studies. The drugs used for this purpose have advantages and disadvantages against each other. Ketamine and propofol have been used most frequently agents and remifentanil is used with increasing frequency in recent years. Investigators will compare ketamine-propofol and ketamine-remifentanyl effects on drug consumption, respiration, hemodynamics and recovery in pediatric colonoscopy patients. Our study is a prospective, randomized comparison of ketamine-propofol and remifentanyl-propofol for sedation and analgesia in pediatric patients during elective colonoscopy. ASA I-II, 2-16 years old, seventy children will included in the study after ethics committee approval and written informed consent from the parents. Children with cardiovascular, cerebral, pulmonary, renal and hepatic diseases will excluded from the study. Patients will be divided into two groups randomly. Patients will fast for at least 6 hours and have an i.v. line in place for the duration of sedation and recovery. All patients will be administered 0,5 mg/kg midazolam orally for premedication 30 minutes before the procedure. Heart rate, systolic and diastolic arterial pressure, peripheral oxygen saturation, respiratory rate and Ramsay sedation scores of all of patients will recorded at baseline, after induction and every 5 minutes during the procedure by the anesthesiologist. All of the patients will receive oxygen (2-4 L/min) through a nasal cannula and 10 ml/kg/h crystalloid infusion perioperatively. The level of recovery at the end of the procedure will be evaluated by Steward Recovery Score.

Group I (RK); 2 mg/kg ketamine and 0,25 µg/kg remifentanyl will be administered for induction in 1 minute. Then 0,1 µg/kg/h remifentanyl infusion will be started.

Group II (PK); 2 mg/kg ketamine and 1 mg/kg propofol will be administered for induction and then 1 mg/kg/h propofol infusion will be started.

In case of movement, crying, heart rate and systolic blood pressure more than 20% increase from baseline; 0.05 to 0.1 mg / kg of remifentanil will be administered in group I, 0.5-1 mg / kg will be administered propofol in group II. Not enough that case 0.5-1 mg / kg of ketamine will be applied.

The anesthesiologist will continue monitoring after completion of colonoscopy until recovery of full consciousness. A Steward recovery score of 7 will be defined as the end of the recovery time. Throughout the process and during the postoperative observation, if systolic blood pressure more than 20% decrease from baseline will be applied 0,1 mg/kg ephedrine, if heart rate more than 20% decrease from baseline 0,01 mg/kg atropine will be applied.Colonoscopy time will be recorded. At the end of the procedure, the gastroenterologist will be asked to give a score in terms of ease attempt. (1=poor, 2=moderate, 3=good, 4=excellent) Adverse events will be recorded, including hypotension (decrease in blood pressure by 20% from baseline), hypertension (increase in blood pressure by 20% from baseline), bradycardia (decrease in heart rate by 20% from baseline), and hypoxia (oxygen desaturation with peripheral oxygen saturation <90%). In addition, the need for additional medication and operator satisfaction among will be compared to the among groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 2-16 years old children

Exclusion Criteria:

* Children with cardiovascular disease,
* Children with cerebral disorder, respiratory disease,
* Children with renal failure
* Children with hepatic failure

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Ketamine, remifentanyl, propofol consumption | 1 hour
  The amount of anesthetic used during colonoscopy will be recorded as milligram/kilogram for each patient.

SECONDARY OUTCOMES:
Blood pressure | 1 hour
  Blood pressure will be followed during colonoscopy and until modified aldrete score will be 9 points.
Hypoxia | 1 hour
  Hypoxia (oxygen desaturation with peripheral oxygen saturation <90%) will be followed during colonoscopy and until modified aldrete score will be 9 points.
Heart rate | 1 hour
  Heart rate will be followed during colonoscopy and until modified aldrete score will be 9 points.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Özcengiz, Prof, Study Chair — Cukurova University; Çağatay Küçükbingöz, Asistant dr, Study Chair — Cukurova University
Locations (1):
- Cukurova University Faculty of Medicine Research Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No